CLINICAL TRIAL: NCT00771368
Title: A Clinical Trial on the Reduction of Bacteria (Including MRSA) in MRSA Positive Ulcers and Lesions
Brief Title: Reduction of Bacteria in MRSA Positive Ulcers
Status: Terminated | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: limited recruitment
Sponsor: Nitric BioTherapeutics, Inc (Industry)
Responsible Party: President & CEO, Nitric BioTherapeutics, Inc.
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CTP 7
Record Dates: First submitted 2008-10-10; First posted 2008-10-13 (Estimated); Last update posted 2012-01-19 (Estimated); Status verified 2012-01

CONDITIONS: Leg Ulcer; Pressure Ulcer
MeSH Terms: conditions — Leg Ulcer; Pressure Ulcer | interventions — Nitric Oxide

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Nitric Oxide (Experimental): gaseous nitric oxide delivered topically for 30 minutes
  Interventions: Drug: Nitric Oxide

INTERVENTIONS:
Drug: Nitric Oxide — 1 % Gaseous Nitric Oxide, delivered for 30 minutes daily for 3 consecutive days

SUMMARY:
The purpose of this study is to determine if gaseous nitric oxide is effective in the treatement of bacteria in MRSA positive ulcers

ELIGIBILITY:
Inclusion Criteria:

* Must have given written informed consent
* Must be 19 years of age or over
* Must have an ulcer or lesion in which the presence of MRSA has been positively identified but which is not clinically infected.
* Must have an Ulcer / Lesion size not to extend beyond the inner borders of the wound cover

Exclusion Criteria:

* Is a female who is pregnant, nursing, or of child bearing potential who is not using an adequate form of contraception (or abstinence)
* Is < 19 years of age
* Has a clinically infected ulcer
* Has an Ulcer / Lesion that is currently treated or has been treated with a topical antimicrobial agent during 3 days prior to enrolment.
* Has been using systemic antibiotics during 7 days prior to enrolment into this study.
* Has an Ulcer / Lesion which is identified as malignant in origin (e.g., Marjolin's ulcer)
* Has an Ulcer / Lesion size beyond the inner borders of the wound cover
* Is septic or has other signs of an invasive infection
* Has used any other investigational product within 30 days preceding study participation.
* Suffers from a condition, which, in the opinion of the Investigator,would compromise his or her safety.
* Suffers from a condition which, in the opinion of the Investigator, would compromise the quality of the data.
* Has a known allergy to any of the products that are part of this protocol
* Suffers from a condition which, in the opinion of the Investigator, would seriously interfere negatively with the normal parameters of immune response to an infection.
* Is using any of the prohibited concomitant medications or treatments

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2009-01; Primary Completion 2009-05 (Actual); Study Completion 2009-06 (Actual)

PRIMARY OUTCOMES:
Reduction in bacteria | Post Treatment Day 3

SECONDARY OUTCOMES:
Incidence of adverse events | 3 days

CONTACTS AND LOCATIONS:
Locations (1):
- Vancouver General Hospital, Vancouver, British Columbia, Canada